CLINICAL TRIAL: NCT07114770
Title: Explore the Impacts of One Session and Multiple Session Theta Burst Stimulation Over Cerebellum in Adults With Autism Spectrum Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202500396A0
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder; Theta Burst Stimulation
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Autistic adults (Experimental): Eligible participants are adults diagnosed with autism who meet the inclusion criteria of the study.
  Interventions: Device: Theta Burst Stimulation (TBS, an advanced variant of repetitive transcranial magnetic stimulation)
- Typically developing adults (Active Comparator): Eligible participants are typically developing adults who meet the study's inclusion criteria.
  Interventions: Device: Theta Burst Stimulation (TBS, an advanced variant of repetitive transcranial magnetic stimulation)

INTERVENTIONS:
Device: Theta Burst Stimulation (TBS, an advanced variant of repetitive transcranial magnetic stimulation) — Participants will receive a single session of either iTBS or cTBS (600 pulses) targeting the right cerebellar Crus I/II. One week after the initial TBS, they will receive another single session of iTBS or cTBS (600 pulses) at the same site.

SUMMARY:
This study aims to establish a personalized theta burst stimulation (TBS, an advanced variant of repetitive transcranial magnetic stimulation, rTMS) protocol considering autistic idiosyncrasy (interindividual variability).

ELIGIBILITY:
Inclusion criteria for autistic adults:

* Autistic adults (≥18 years old), confirmed by Autism Diagnostic Observation Schedule.
* DSM-5 severity level of ASD: level 1 or level 2

Inclusion criteria for typically developing control:

* ≥18 years old without autism spectrum disorder

Exclusion criteria for all participants:

* Previous or current severe neurological disorders, especially epilepsy
* Previous or current severe systemic diseases such as cardiovascular disease, diabetes or hypertension
* Previous or current severe brain injury
* Implementation of metal materials such as a pacemaker or medication pump
* Previous or current severe psychiatric disorders such as schizophrenia, bipolar disorder, severe major depressive disorder or substance abuse
* Pregnancy
* Intracranial space occupied lesions
* Previous brain surgery or central nerve system infection
* Concurrent use of medications which increased the risk of seizure attack
* Participate in another clinical trial within one month
* With damaged skin at the stimulated region
* With multiple sclerosis
* With large ischemic scars
* Have experienced sleep disorders during brain stimulation
* Severe alcoholism
* Concurrent use of antiepileptic drugs
* Uncontrollable migraines due to increased intracranial pressure
* Unsuitable for MRI (e.g. those with claustrophobia)
* Unsuitable for EEG
* DSM-5 severity level of ASD: level 3
* Suicidal ideation within one year

Withdrawal criteria:

* Seizure attack during the study period
* Autistic symptoms worsened obviously during the study period (change of DSM-5 severity level)
* Extreme agitation or irritability during the study period
* Participants request
* Clinical symptoms worsened obviously during study period
* Start to use antiepileptic drugs during study period
* Suicidal ideation or self-harm behaviors during study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional MRI (default mode network) - BOLD Signal | Baseline, Week 1, Week 2
  Blood-oxygen-level-dependent (BOLD) signal is a measurement used in fMRI, which reflects the neural activity.
MEP amplitude | Baseline
  MEP (motor evoked potential) amplitude is a measure of corticospinal excitability.
MEP amplitude | Week 1 (5 minutes post-TBS)
  MEP (motor evoked potential) amplitude is a measure of corticospinal excitability.
MEP amplitude | Week 2 (5 minutes post-TBS)
  MEP (motor evoked potential) amplitude is a measure of corticospinal excitability.
MEP amplitude | Week 1 (10 minutes post-TBS)
  MEP (motor evoked potential) amplitude is a measure of corticospinal excitability.
MEP amplitude | Week 2 (10 minutes post-TBS)
  MEP (motor evoked potential) amplitude is a measure of corticospinal excitability.
MEP amplitude | Week 1 (15 minutes post-TBS)
  MEP (motor evoked potential) amplitude is a measure of corticospinal excitability.
MEP amplitude | Week 2 (15 minutes post-TBS)
  MEP (motor evoked potential) amplitude is a measure of corticospinal excitability.
MEP amplitude | Week 1 (20 minutes post-TBS)
  MEP (motor evoked potential) amplitude is a measure of corticospinal excitability.
MEP amplitude | Week 2 (20 minutes post-TBS)
  MEP (motor evoked potential) amplitude is a measure of corticospinal excitability.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan